CLINICAL TRIAL: NCT06695793
Title: Niche Investigated: Closure of Hysterotomy & Evaluation of 3 Suturing Techniques (Running, Interrupted, and Locked)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdalla Mousa, Lecturer of obgyn Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-308-2024
Record Dates: First submitted 2024-11-17; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Caesarean Scar Niche

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A) (Experimental): Interrupted Sutures: The first layer of the uterine incision will be closed using individual, separate sutures placed at regular intervals along the incision line. Each suture will be tied independently, ensuring adequate apposition of uterine tissue, followed by a second layer of running continuous sutures.
  Interventions: Procedure: Interrupted Sutures
- Group (B) (Experimental): Locked Sutures: The first layer of the uterine incision will be closed using continuous sutures placed along the uterine incision, incorporating a locking technique at specified intervals to prevent unraveling. The knots will be securely tied to maintain tissue approximation, followed by a second layer of running continuous sutures.
  Interventions: Procedure: Locked Sutures
- Group (C) (Experimental): Running Continuous Sutures: Double layer closure of uterine incision using running continuous suture used to close the uterine incision without interruption, providing seamless tissue approximation throughout the incision length.
  Interventions: Biological: Running Continuous Sutures

INTERVENTIONS:
Procedure: Interrupted Sutures — The first layer of uterine incision will be closed using individual, separate sutures placed at regular intervals along the incision line. Each suture will be tied independently, ensuring adequate apposition of uterine tissue, followed by a second layer of running continuous sutures.
  Arms: Group (A)
Procedure: Locked Sutures — The first layer of uterine incision will be closed using continuous sutures placed along the uterine incision, incorporating a locking technique at specified intervals to prevent unraveling. The knots will be securely tied to maintain tissue approximation, followed by a second layer of running continuous sutures.
  Arms: Group (B)
Biological: Running Continuous Sutures — Double layer closure of uterine incision using running continuous suture used to close the uterine incision without interruption, providing seamless tissue approximation throughout the incision length.
  Arms: Group (C)

SUMMARY:
This study aims to explore the impact of three different suturing techniques (Running, Interrupted & Locked) that used to close the uterine incision at the cesarean section on the formation of a cesarean scar niche

ELIGIBILITY:
Inclusion Criteria:

1. Women with a singleton pregnancy scheduled for elective cesarean section
2. Gestational age at the time of cesarean section between 38 and 40 weeks.
3. Willingness to participate in the study and provide informed consent
4. Age between 18 and 35 years old.
5. BMI <30

Exclusion Criteria:

1. Known uterine anomalies or previous uterine surgery (e.g, myomectomy, uterine septum resection)
2. Pre-existing medical conditions contraindicating cesarean delivery or affecting uterine healing (e.g., Anemia, Diabetes)
3. Current smokers.
4. Non-cephalic presentation of the fetus.
5. Low-lying anterior wall placenta and placenta previa.
6. Inability to provide informed consent (e.g., cognitive impairment, language barrier)
7. Any condition deemed by the attending physician to pose a risk to the participant or compromise the study's integrity, for example, Patients who will require excessive suturing for further hemostasis or those who require ligation of one or both uterine arteries

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Presence of caesarean scar niche and its dimensions. | 6-12 weeks post-cesarean section
  Follow-up visits will be scheduled at 6-12 weeks post-cesarean section to assess caesarean section niche formation using trans-vaginal ultrasound using Samsung Elite with endovaginal probe of frequency 6 - 12 MHz. Trained sonographers, blinded to the participants' suturing group, will perform the ultrasound examinations to evaluate caesarean section niche presence and its dimensions.

SECONDARY OUTCOMES:
Operative time | during operation
Estimate blood loss | during operation

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt